CLINICAL TRIAL: NCT02545192
Title: A Pilot Study of Low Field Magnetic Stimulation in PTSD: Three Daily Treatments
Acronym: LFMS in PTSD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Michael Rohan, Imaging Physicist, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015P001621
Record Dates: First submitted 2015-08-06; First posted 2015-09-09 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active LFMS treatment (Experimental): 20 minutes of active Low Field Magnetic Stimulation using the LFMS device.
  Interventions: Device: Low Field Magnetic Stimulation
- Sham LFMS treatment (Sham Comparator): 20 minutes of sham Low Field Magnetic Stimulation using the LFMS device.
  Interventions: Device: Low Field Magnetic Stimulation

INTERVENTIONS:
Device: Low Field Magnetic Stimulation — The LFMS Device is an electromagnetic coil situated on a cylinder with an inside diameter of 13.2 inches. It produces weak electromagnetic fields at a frequency of about 1000Hz; the magnetic fields are less than 30 Gauss and the electric fields are up to 1.43 V/m. A fully detailed description of the electromagnetic field distribution and waveform has been presented in the IDE submission to the FDA (and determined to be a non-significant risk device).
  Other Names: LFMS

SUMMARY:
The investigators propose to make the first observations of LFMS treating a population of subjects with PTSD. A positive outcome for this study could translate directly into a new treatment modality for symptoms of PTSD in both acute and chronic situations. The investigator's goal is to demonstrate the safety and efficacy of LFMS as a possible aid in the treatment of PTSD.

DETAILED DESCRIPTION:
The Low Field Magnetic Stimulation (LFMS) procedure is an application of a series of electromagnetic pulses to the brain lasting twenty minutes. The field and timing parameters of the LFMS pulses, such as pulse timing, duration, frequency, and electric and magnetic field distribution and direction are different from other neurostimulation methods. LFMS electromagnetic fields are significantly weaker than those occurring in electroconvulsive therapy (ECT) and repeated transcranial magnetic stimulation (rTMS).

LFMS was discovered at McLean Hospital and has been studied as an experimental antidepressant treatment at McLean. Results from the investigator's single-visit protocol (2006-P-001655) are encouraging, and demonstrate an immediate mood improvement from LFMS in depressed subjects. This indicates that LFMS continues to show potential as a treatment for depression. The profile of clinical response to LFMS that was observed in that study included improvement in symptoms of anxiety. In this current proposal the investigator's will study the effects of LFMS on these symptoms of depression and anxiety that are present in a population with a primary diagnosis of PTSD. The proposed protocol involves three treatments on consecutive days with follow-up ratings one week after the first treatment and follow-up by phone ratings in weeks three and four after the first treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be men or women between the ages of 21-65.
2. Subjects will meet Diagnostics and Statistical Manual of Mental Disorders (DSM-IV) criteria for Post Traumatic Stress Disorder (PTSD), current.
3. Subject must have a PTSD Check List-5 (PCL-5) score greater than 38.
4. Subjects must be capable of providing informed consent.
5. Subjects must have an established residence and phone.
6. Subjects may be medicated or unmedicated.

Exclusion Criteria:

1. Dangerous or active suicidal ideation.
2. Pregnant or planning on becoming pregnant.
3. Substance abuse (cannot meet DSM criteria for substance abuse, no significant drug abuse within last 3 months, no major polysubstance abuse history, no history of dependence in last year, no drug use within last month).
4. Significant medical or neurological illness that might pose a risk to study enrollment or interfere with interpretation of study data.
5. Subjects must not have serious physical illnesses, neurological diseases or dementias.
6. Changes in psychiatric medication (e.g. dose or drug) within 6 weeks prior to enrollment.
7. History of an Axis 2 disorder, schizophrenia or schizoaffective disorder.
8. Contraindications for magnetic resonance imaging (MRI): Presence of a pacemaker, neurostimulator, or metal in head or neck.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change in depression | 1 week
  Change in depression as measured by the Montgomery Asberg Depression Rating Scale in subjects receiving active LFMS treatment relative to sham treatment
Change in anxiety | 1 week
  Change in anxiety levels as measured by the Hamilton Anxiety Rating Scale in subjects receiving active LFMS treatment relative to sham treatment

SECONDARY OUTCOMES:
Improvement in core PTSD symptoms | 1 week
  Measures of core PTSD symptoms will show improvement over one week in subjects receiving active LFMS treatment relative to sham treatment
Daily improvements in short-term measures of depression | 24 hrs
  Short term measures of depression will show improvements in subjects receiving active LFMS treatment relative to sham treatment
Daily improvements in short-term measures of anxiety | 24 hrs
  Short term measures of anxiety will show improvements in subjects receiving active LFMS treatment relative to sham treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Rohan, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Rohan M, Parow A, Stoll AL, Demopulos C, Friedman S, Dager S, Hennen J, Cohen BM, Renshaw PF. Low-field magnetic stimulation in bipolar depression using an MRI-based stimulator. Am J Psychiatry. 2004 Jan;161(1):93-8. doi: 10.1176/appi.ajp.161.1.93. PMID 14702256
- [Result] Rohan ML, Yamamoto RT, Ravichandran CT, Cayetano KR, Morales OG, Olson DP, Vitaliano G, Paul SM, Cohen BM. Rapid mood-elevating effects of low field magnetic stimulation in depression. Biol Psychiatry. 2014 Aug 1;76(3):186-93. doi: 10.1016/j.biopsych.2013.10.024. Epub 2013 Nov 12. PMID 24331545